CLINICAL TRIAL: NCT02367287
Title: Assessing the Impact of Diet on Inflammation in Healthy and Obese Adults in a Cross-Sectional Phenotyping Study
Brief Title: USDA Western Human Nutrition Research Center (WHNRC) Cross-Sectional Nutritional Phenotyping Study
Status: Completed | Type: Observational
Sponsor: USDA, Western Human Nutrition Research Center (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 691654; 2032-53000-001-00 (Other Grant/Funding Number: United States Department of Agriculture)
Record Dates: First submitted 2015-02-12; First posted 2015-02-20 (Estimated); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Obesity; Inflammation
Keywords: Diet; Phenotype; Immunology; Microbiota; Metabolomics; Physical activity; Neuroendocrine system; Nutritional Physiological Phenomena
MeSH Terms: conditions — Obesity; Inflammation; Motor Activity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Whole blood, stool
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Sampling strata: Stratified analyses of primary and secondary outcomes based on variables of interest (e.g. sex, age, or BMI) may occur prior to achieving the target for total study enrollment.

SUMMARY:
Although the diet of the US population meets or exceeds recommended intake levels of most essential nutrients, the quality of the diet consumed by many Americans is sub-optimal due to excessive intake of added sugars, solid fats, refined grains, and sodium. The foundations and outcomes of healthy vs. unhealthy eating habits and activity levels are complex and involve interactions between the environment and innate physiologic/genetic background. For instance, emerging research implicates chronic and acute stress responses and perturbations in the Hypothalamic-Pituitary-Adrenal axis in triggering obesity-promoting metabolic changes and poor food choices. In addition, the development of many chronic diseases, including cardiovascular disease, diabetes, cancer, asthma and autoimmune disease, results from an overactive immune response to host tissue or environmental antigens (e.g. inhaled allergens). A greater understanding is needed of the distribution of key environment-physiology interactions that drive overconsumption, create positive energy balance, and put health at risk.

Researchers from the United States Department of Agriculture (USDA) Western Human Nutrition Research Center are conducting a cross-sectional "metabolic phenotyping" study of healthy people in the general population. Observational measurements include the interactions of habitual diet with the metabolic response to food intake, production of key hormones, the conversion of food into energy: the metabolism of fats, proteins, and carbohydrates, characteristics of the immune system, stress response, gut microbiota (bacteria in the intestinal tract), and cardiovascular health. Most outcomes will be measured in response to a mixed macronutrient/high fat challenge meal.

DETAILED DESCRIPTION:
Many inflammatory responses can be modulated by specific dietary components. For example, in cardiovascular disease, macrophages and T-cells react with oxidized LDL (an endogenous modified antigen) to produce arterial plaque and subsequent blockage of coronary arteries. High intake of saturated fats (or simple sugars that drive synthesis of saturated fatty acids) may promote this inflammation by affecting macrophages and T-cells. Conversely, increased intake of omega-3 fatty acids may decrease inflammation by suppression of macrophage and T-cell pro-inflammatory activity. Long-term sub-clinical inflammation caused by intestinal bacteria has been linked to the development of Irritable Bowel Disease and related disorders. Low intake of fruits, vegetables, or whole grains or high intake of saturated fats may promote sub-clinical gut inflammation by promoting dysbiosis of the gut microbiota. Allergic asthma develops in predisposed individuals as a result of an overactive allergic-type immune response to inhaled environmental allergens. Dietary factors such as vitamin D and omega-3 fatty acids may diminish pro-inflammatory responses to environmental allergens by promoting the development of T-regulatory cells and other anti-inflammatory factors.

Individual variability in chronic disease risk is well recognized. For example, why does excess adiposity lead to disease in some individuals and not others? The nature of the fat tissue rather than the abundance, may impact cross-talk with other metabolically-relevant tissues and affect disease risk. It is important to characterize healthy vs. unhealthy phenotypes across various tissues and to understand how micro- and macro-nutrients interact with molecular and metabolic pathways to support a healthy body weight. This study brings together scientists with expertise in nutritional sciences, immunology, analytical chemistry, physiology, neuroendocrinology, and behavior to understand how diet impacts metabolism and disease risk through the interplay and coordination of signals and metabolites arising from multiple organ systems.

The overall objective is to characterize the phenotypic profile of participants according to their immunologic, physiologic, neuroendocrine, and metabolic responses to a dietary challenge and a physical fitness challenge by addressing the specific aims listed below. The cross-sectional study is organized into two study visits (Visit 1 and Visit 2) separated by approximately two weeks of at-home specimen and data collection.

Specific Aim 1: To determine if diet quality is independently associated with systemic immune activation, inflammation, or oxidative stress differentiated by:

1. pro-inflammatory T-helper cells (Th1, Th2, and Th17 cells) and related cytokines
2. anti-inflammatory T-regulatory cells and related cytokines
3. dysbiosis of the gut microbiota and markers of gut inflammation (e.g. neopterin and myeloperoxidase)

   a. and to evaluate the association between dysbiosis of the gut microbiota, gut inflammation, and systemic immune activation
4. plasma metabolomic response to a mixed macronutrient challenge meal (includes diet quality and physical activity as independent variables)
5. endothelial (dys)function and vascular reactivity

Specific Aim 2: To determine if a high fat/sugar challenge meal induces differential effects over time (0-6h postprandial) according to habitual diet characteristics, physical activity levels, stress levels, age, sex, or BMI on:

1. postprandial monocyte activation
2. plasma lipid metabolomic responses including non-esterified fatty acids, phospholipids, triacylglycerols, red blood cell fatty acids, endocannabinoids, bile acids, eicosanoids and related oxylipins, ceramides, sphingoid bases, and acylcarnitines
3. plasma amino acid metabolomics
4. glucose metabolism and metabolic flexibility (i.e. the ability to switch from glucose to lipid oxidation as energy sources)
5. changes in endocrinology and self-report of hunger and satiety
6. postprandial free cortisol

Specific Aim 3: To determine the mechanisms of:

1. postprandial monocyte activation
2. suppression of challenge-meal induced monocyte activation by docosahexaenoic acid (DHA) (in an ex vivo experiment using a subset of samples)

Specific Aim 4: To evaluate the associations between eating behavior, physical activity, and/or anthropometry and the outcomes:

1. endocrinology of hunger and satiety
2. plasma metabolomic responses
3. vulnerability and resistance to stress
4. endothelial (dys)function and vascular reactivity
5. prediction of insulin sensitivity

Specific Aim 5: To determine how genetic variants affect nutrient metabolism, cardiovascular physiology, and immune function and improve understanding of how dietary factors affect these metabolic, cardiovascular and immune phenotypes.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 y
* Male or female
* Body Mass Index 18.5-45.0 kg/m2 (Normal to obese)

Exclusion Criteria:

* Pregnant or lactating women
* Known allergy to egg-white protein
* Systolic blood pressure greater than 140 mm Hg or diastolic blood pressure greater than 90 mm Hg measured on three separate occasions
* Diagnosed active chronic diseases for which the individual is currently taking daily medication, including but not limited to:

  * Diabetes mellitus
  * Cardiovascular disease
  * Cancer
  * Gastrointestinal disorders
  * Kidney disease
  * Liver disease
  * Bleeding disorders
  * Asthma
  * Autoimmune disorders
  * Hypertension
  * Osteoporosis
* Recent minor surgery (within 4 wk) or major surgery (within 16 wk)
* Recent antibiotic therapy (within 4 wk)
* Recent hospitalization (within 4 wk)
* Use of prescription medications at the time of the study that directly affect endpoints of interest (e.g. hyperlipidemia, glycemic control, steroids, statins, anti-inflammatory agents, and over-the-counter weight loss aids)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy people in the general population
Sampling Method: Non-Probability Sample
Enrollment: 393 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2019-07-24 (Actual); Study Completion 2019-07-24 (Actual)

PRIMARY OUTCOMES:
Baseline level and change in systemic immune activation following challenge meal | 0, 0.5, 3, and 6 hours postprandial
  Number and activation level of pro-inflammatory T-helper (Th) cells (Th1, Th2 and Th17), T-regulatory (Treg) cells, and B cells will be measured in fasting blood. Monocytes and neutrophils will be measured in fasting and postprandial blood.
Baseline level and change in plasma metabolome | 0, 0.5, 3, and 6 hours postprandial
  Plasma fatty acid profiles of non-esterified fatty acids, phospholipids, triacylglycerols, red blood cell fatty acids, endocannabinoids, bile acids, eicosanoids and related oxylipins, ceramides, sphingoid bases, acylcarnitines, amino acids and other metabolites measured in response to a challenge meal.

SECONDARY OUTCOMES:
Baseline level and change in glucose metabolism | 0, 0.5, 3, and 6 hours postprandial
  Glucose and insulin measured in response to a challenge meal.
Baseline level and change in appetitive hormones | 0, 0.5, 3, and 6 hours postprandial
  Cholecystokinin, incretins, Peptide YY 3-36, ghrelin measured in response to a challenge meal.
Baseline level and change in mitogen activated protein (MAP) kinase activity | 0, 0.5, 3 and 6 hours postprandial
  Mononuclear cells or B cells will be measured for MAP kinase activities in fasting and postprandial blood.
Baseline level and change in dietary-responsive, circulating microRNA | 0, 0.5, 3, and 6 hours postprandial
  Plasma microRNA measured in response to a challenge meal
Baseline level and change in RNA transcriptome | 0, 3, and 6 hours postprandial
  Transcriptome RNA sequenced in whole blood
Genome Wide Association Study (GWAS) | 0 hours (fasting)
  DNA sequence from whole blood will be analyzed
General health | 0 hours (Fasting)
  Clinical chemistry panel and complete blood count
Anthropometrics | single time point
  Height (cm), weight (kg), waist and hip circumference (cm)
Vital signs | single time point
  Blood pressure (mmHg), pulse rate (beats per minute) and temperature (degrees F).
Body composition | single time point
  Body composition (percent body fat) and bone mineral density by Dual energy X-ray Absorptiometry scan.
Resting and change in metabolism | 0, 0.5, 3, and 6 hours postprandial
  Resting and postprandial metabolic rates, including respiratory exchange ratios.
Gut microbiota | single time point
  Gut microbiota composition and gene content will be assessed in stool using polymerase chain reaction (PCR) and sequencing
Gut microbiota fermentation capacity | single time point
  The fermentation capacity of microbiota will be measured from a single stool sample
Gut microbiota pathogen resistance capacity | single time point
  The pathogen resistance capability of microbiota will be measured from a single stool sample
Gut inflammation | single time point
  Gut inflammation will be assessed by measuring molecules in stool and/or the response of intestinal epithelial cell cultures to fecal waters from a single stool sample.
Stool metabolites | single time point
  Volatile and short chain fatty acids and bile acids will be measured in a single stool sample.
Stool RNA markers | single time point
  RNA markers will provide a measure of genes expressed by cells of the colon naturally present in a single stool sample
Baseline and change in hunger and appetite | 0, 1, 2, 3, 4, 5, and 6 hours postprandial
  Perceived hunger and fullness will be measured using a visual analog scale. Responses will be a marked on an unsegmented line from 0 or "not at all" to 5 or "extremely."
Baseline and change in gut fermentation profile | 0, 1, 2, 3, 4, 5, and 6 hours postprandial
  Breath hydrogen and methane measured in response to a challenge meal.
Recent dietary intake | Three 24-hour dietary recalls collected at home
  Random selection of 2 week days and 1 weekend day for 24-hour recall using an automated multi-pass method
Dietary intake | single time point
  Food frequency questionnaire (FFQ)
Behavior assessment | single time point
  Chronic stress questionnaire, food choice questionnaires, and a food preference activity.
Taste thresholds | single time point
  Sampling tastes of sweet, salty, and bitter solutions in comparison to water to determine threshold of taste detection.
Skin reflectance | single time point
  Spectrophotometric measure of skin pigmentation for assessment of vitamin D status.
Peripheral arterial tone | single time point
  Use of the EndoPAT system to measure blood vessel tone.
Pulmonary function | single time point
  Forced expiratory lung volume test
Pulmonary inflammation | single time point
  Pulmonary inflammation measured as exhaled nitric oxide (NO)
Executive function | single time point
  Executive function will be assessed using Cambridge Neuropsychological Test Automated Battery (CANTAB) and Iowa Gambling Task
Cognitive function | single time point
  Measured by Wechsler Abbreviated Standard Intelligence test.
Aerobic fitness assessment | single time point
  Pulse rate (bpm) and recovery after a 3 min YMCA Step Test
Submaximal oxygen consumption | single time point
  The submaximal volume of oxygen consumed during a 4 minute treadmill walking protocol (VO2max) (ml/kg*min)
Physical activity | daily, for 7 days
  Use of an accelerometer worn on the hip for 7 days
Usual physical activity | single time point
  Activity recall using a questionnaire
Heart rate variability and autonomic nerve conductivity | single time point
  Monitoring of autonomic balance, cardiac performance, and respiratory measurements and activity using MindWare Mobile Impedance Cardiograph.
Allostatic Load | single time point
  An aggregate score derived from measures of urinary cortisol, norepinephrine, epinephrine, blood cholesterol, high sensitivity c-reactive protein, and hemoglobin A1C.
Baseline and change in salivary cortisol in response to test meal | 0, immediately post-prandial, 30, 60, and 90 minutes post-prandial
  Salivary cortisol measured by enzyme-linked immunosorbent assay (ELISA)
Baseline and change in salivary cortisol in response to exercise | 0, immediately post-exercise, 30, 60, and 90 minutes post-exercise
  Salivary cortisol measured by enzyme-linked immunosorbent assay (ELISA)
Baseline and change in salivary cortisol in response to emotional recall task | 0, immediately post-task, 30, 60, and 90 minutes post-task
  Salivary cortisol measured by enzyme-linked immunosorbent assay (ELISA)
Baseline and change in breath aldehydes | 0, 1, 4 and 6 hours postprandial
  The concentration of aldehydes present in human breath before and after a high-fat meal will be measured by mass spectrometry

CONTACTS AND LOCATIONS:
Overall Officials: Charles B Stephensen, Ph.D., Principal Investigator — USDA, Western Human Nutrition Research Center; Brian J Bennett, Ph.D., Principal Investigator — USDA, Western Human Nutrition Research Center
Locations (1):
- USDA, Western Human Nutrition Research Center, Davis, California, United States

REFERENCES:
- [Background] Wopereis S, Wolvers D, van Erk M, Gribnau M, Kremer B, van Dorsten FA, Boelsma E, Garczarek U, Cnubben N, Frenken L, van der Logt P, Hendriks HF, Albers R, van Duynhoven J, van Ommen B, Jacobs DM. Assessment of inflammatory resilience in healthy subjects using dietary lipid and glucose challenges. BMC Med Genomics. 2013 Oct 27;6:44. doi: 10.1186/1755-8794-6-44. PMID 24160467
- [Background] Pellis L, van Erk MJ, van Ommen B, Bakker GC, Hendriks HF, Cnubben NH, Kleemann R, van Someren EP, Bobeldijk I, Rubingh CM, Wopereis S. Plasma metabolomics and proteomics profiling after a postprandial challenge reveal subtle diet effects on human metabolic status. Metabolomics. 2012 Apr;8(2):347-359. doi: 10.1007/s11306-011-0320-5. Epub 2011 May 28. PMID 22448156
- [Background] Krug S, Kastenmuller G, Stuckler F, Rist MJ, Skurk T, Sailer M, Raffler J, Romisch-Margl W, Adamski J, Prehn C, Frank T, Engel KH, Hofmann T, Luy B, Zimmermann R, Moritz F, Schmitt-Kopplin P, Krumsiek J, Kremer W, Huber F, Oeh U, Theis FJ, Szymczak W, Hauner H, Suhre K, Daniel H. The dynamic range of the human metabolome revealed by challenges. FASEB J. 2012 Jun;26(6):2607-19. doi: 10.1096/fj.11-198093. Epub 2012 Mar 16. PMID 22426117
- [Background] Robles Alonso V, Guarner F. Linking the gut microbiota to human health. Br J Nutr. 2013 Jan;109 Suppl 2:S21-6. doi: 10.1017/S0007114512005235. PMID 23360877
- [Background] Baldiviez LM, Keim NL, Laugero KD, Hwang DH, Huang L, Woodhouse LR, Burnett DJ, Zerofsky MS, Bonnel EL, Allen LH, Newman JW, Stephensen CB. Design and implementation of a cross-sectional nutritional phenotyping study in healthy US adults. BMC Nutr. 2017 Oct 19;3:79. doi: 10.1186/s40795-017-0197-4. eCollection 2017. PMID 32153856
- [Result] Oliver A, Alkan Z, Stephensen CB, Newman JW, Kable ME, Lemay DG. Diet, Microbiome, and Inflammation Predictors of Fecal and Plasma Short-Chain Fatty Acids in Humans. J Nutr. 2024 Nov;154(11):3298-3311. doi: 10.1016/j.tjnut.2024.08.012. Epub 2024 Aug 20. PMID 39173973
- [Result] James KL, Gertz ER, Kirschke CP, Allayee H, Huang L, Kable ME, Newman JW, Stephensen CB, Bennett BJ. Trimethylamine N-Oxide Response to a Mixed Macronutrient Tolerance Test in a Cohort of Healthy United States Adults. Int J Mol Sci. 2023 Jan 20;24(3):2074. doi: 10.3390/ijms24032074. PMID 36768394
- [Result] Riazati N, Kable ME, Newman JW, Adkins Y, Freytag T, Jiang X, Stephensen CB. Associations of microbial and indoleamine-2,3-dioxygenase-derived tryptophan metabolites with immune activation in healthy adults. Front Immunol. 2022 Sep 29;13:917966. doi: 10.3389/fimmu.2022.917966. eCollection 2022. PMID 36248784
- [Result] Chin EL, Huang L, Bouzid YY, Kirschke CP, Durbin-Johnson B, Baldiviez LM, Bonnel EL, Keim NL, Korf I, Stephensen CB, Lemay DG. Association of Lactase Persistence Genotypes (rs4988235) and Ethnicity with Dairy Intake in a Healthy U.S. Population. Nutrients. 2019 Aug 10;11(8):1860. doi: 10.3390/nu11081860. PMID 31405126
- [Result] Bouzid YY, Arsenault JE, Bonnel EL, Cervantes E, Kan A, Keim NL, Lemay DG, Stephensen CB. Effect of Manual Data Cleaning on Nutrient Intakes Using the Automated Self-Administered 24-Hour Dietary Assessment Tool (ASA24). Curr Dev Nutr. 2021 Feb 2;5(3):nzab005. doi: 10.1093/cdn/nzab005. eCollection 2021 Mar. PMID 33763626
- [Result] Lemay DG, Baldiviez LM, Chin EL, Spearman SS, Cervantes E, Woodhouse LR, Keim NL, Stephensen CB, Laugero KD. Technician-Scored Stool Consistency Spans the Full Range of the Bristol Scale in a Healthy US Population and Differs by Diet and Chronic Stress Load. J Nutr. 2021 Jun 1;151(6):1443-1452. doi: 10.1093/jn/nxab019. PMID 33704458
- [Derived] Blecksmith SE, Oliver A, Alkan Z, Lemay DG. Gut Microbiome Genes Involved in Plant and Mucin Breakdown Correlate with Diet and Gastrointestinal Inflammation in Healthy United States Adults. J Nutr. 2025 Nov;155(11):3757-3768. doi: 10.1016/j.tjnut.2025.08.027. Epub 2025 Sep 1. PMID 40902732
- [Derived] Stephensen CB, Jiang X, Gale B, Peerson JM. Association of Healthy Eating Index-2015 Total and Component Scores with Measures of Inflammation and Immune Activation in Healthy Adults. J Nutr. 2025 Mar;155(3):994-1004. doi: 10.1016/j.tjnut.2025.01.005. Epub 2025 Jan 7. PMID 39788323
- [Derived] Riazati N, Engle-Stone R, Stephensen CB. Association of Vitamin D Status with Immune Markers in a Cohort of Healthy Adults. J Nutr. 2025 Feb;155(2):621-633. doi: 10.1016/j.tjnut.2024.12.010. Epub 2024 Dec 21. PMID 39716659
- [Derived] Wilson SM, Oliver A, Larke JA, Naveja JJ, Alkan Z, Awika JM, Stephensen CB, Lemay DG. Fine-Scale Dietary Polyphenol Intake Is Associated with Systemic and Gastrointestinal Inflammation in Healthy Adults. J Nutr. 2024 Nov;154(11):3286-3297. doi: 10.1016/j.tjnut.2024.08.010. Epub 2024 Aug 18. PMID 39163972
- [Derived] Bouzid YY, Wilson SM, Alkan Z, Stephensen CB, Lemay DG. Lower Diet Quality Associated with Subclinical Gastrointestinal Inflammation in Healthy United States Adults. J Nutr. 2024 Apr;154(4):1449-1460. doi: 10.1016/j.tjnut.2024.02.030. Epub 2024 Mar 1. PMID 38432562
- [Derived] Kable ME, Chin EL, Huang L, Stephensen CB, Lemay DG. Association of Estimated Daily Lactose Consumption, Lactase Persistence Genotype (rs4988235), and Gut Microbiota in Healthy Adults in the United States. J Nutr. 2023 Aug;153(8):2163-2173. doi: 10.1016/j.tjnut.2023.06.025. Epub 2023 Jun 23. PMID 37354976
- [Derived] Snodgrass RG, Jiang X, Stephensen CB, Laugero KD. Cumulative physiological stress is associated with age-related changes to peripheral T lymphocyte subsets in healthy humans. Immun Ageing. 2023 Jun 23;20(1):29. doi: 10.1186/s12979-023-00357-5. PMID 37353855
- [Derived] Larke JA, Bacalzo N, Castillo JJ, Couture G, Chen Y, Xue Z, Alkan Z, Kable ME, Lebrilla CB, Stephensen CB, Lemay DG. Dietary Intake of Monosaccharides from Foods is Associated with Characteristics of the Gut Microbiota and Gastrointestinal Inflammation in Healthy US Adults. J Nutr. 2023 Jan;153(1):106-119. doi: 10.1016/j.tjnut.2022.12.008. Epub 2022 Dec 26. PMID 36913444
- [Derived] Snodgrass RG, Jiang X, Stephensen CB. Monocyte subsets display age-dependent alterations at fasting and undergo non-age-dependent changes following consumption of a meal. Immun Ageing. 2022 Sep 14;19(1):41. doi: 10.1186/s12979-022-00297-6. PMID 36104734
- [Derived] Wang YE, Kirschke CP, Woodhouse LR, Bonnel EL, Stephensen CB, Bennett BJ, Newman JW, Keim NL, Huang L. SNPs in apolipoproteins contribute to sex-dependent differences in blood lipids before and after a high-fat dietary challenge in healthy U.S. adults. BMC Nutr. 2022 Sep 1;8(1):95. doi: 10.1186/s40795-022-00592-x. PMID 36050800
- [Derived] Newman JW, Krishnan S, Borkowski K, Adams SH, Stephensen CB, Keim NL. Assessing Insulin Sensitivity and Postprandial Triglyceridemic Response Phenotypes With a Mixed Macronutrient Tolerance Test. Front Nutr. 2022 May 11;9:877696. doi: 10.3389/fnut.2022.877696. eCollection 2022. PMID 35634390
- [Derived] Oliver A, Xue Z, Villanueva YT, Durbin-Johnson B, Alkan Z, Taft DH, Liu J, Korf I, Laugero KD, Stephensen CB, Mills DA, Kable ME, Lemay DG. Association of Diet and Antimicrobial Resistance in Healthy U.S. Adults. mBio. 2022 Jun 28;13(3):e0010122. doi: 10.1128/mbio.00101-22. Epub 2022 May 10. PMID 35536006
- [Derived] Kable ME, Chin EL, Storms D, Lemay DG, Stephensen CB. Tree-Based Analysis of Dietary Diversity Captures Associations Between Fiber Intake and Gut Microbiota Composition in a Healthy US Adult Cohort. J Nutr. 2022 Mar 3;152(3):779-788. doi: 10.1093/jn/nxab430. PMID 34958387
- [Derived] Chin EL, Van Loan M, Spearman SS, Bonnel EL, Laugero KD, Stephensen CB, Lemay DG. Machine Learning Identifies Stool pH as a Predictor of Bone Mineral Density in Healthy Multiethnic US Adults. J Nutr. 2021 Nov 2;151(11):3379-3390. doi: 10.1093/jn/nxab266. PMID 34313764
- [Derived] Artegoitia VM, Krishnan S, Bonnel EL, Stephensen CB, Keim NL, Newman JW. Healthy eating index patterns in adults by sex and age predict cardiometabolic risk factors in a cross-sectional study. BMC Nutr. 2021 Jun 22;7(1):30. doi: 10.1186/s40795-021-00432-4. PMID 34154665
- [Derived] Mo Z, Huang S, Burnett DJ, Rutledge JC, Hwang DH. Endotoxin May Not Be the Major Cause of Postprandial Inflammation in Adults Who Consume a Single High-Fat or Moderately High-Fat Meal. J Nutr. 2020 May 1;150(5):1303-1312. doi: 10.1093/jn/nxaa003. PMID 32040591
- See also: WHNRC recruiting website — http://www.ars.usda.gov/Main/docs.htm?docid=11240